CLINICAL TRIAL: NCT07249307
Title: Study on Key Technologies for High-throughput Large-model-based AI-assisted Diagnosis Using OCT
Brief Title: High-throughput Large-model-based AI-assisted Diagnosis Using OCT
Status: Not yet recruiting | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: K9164
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Diabetic Retinopathy (DR); Retinal Vein Occlusion (RVO); Age-Related Macular Degeneration (AMD); Pathologic Myopia; Glaucoma
MeSH Terms: conditions — Diabetic Retinopathy; Retinal Vein Occlusion; Macular Degeneration; Glaucoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Diabetic Retinopathy Cohort: Patients undergoing routine OCT/OCTA examinations with clinically diagnosed diabetic retinopathy.
  Interventions: Other: No intervention
- Branch Retinal Vein Occlusion Cohort: Patients with BRVO receiving standard clinical imaging evaluation.
  Interventions: Other: No intervention
- Central Retinal Vein Occlusion Cohort: Patients with CRVO undergoing OCT/OCTA imaging as part of routine care.
  Interventions: Other: No intervention
- Age-related Macular Degeneration Cohort: Patients diagnosed with AMD and evaluated using OCT/OCTA.
  Interventions: Other: No intervention
- Pathologic Myopia with Choroidal Neovascularization Cohort: Patients with pathologic myopia and CNV who undergo OCT/OCTA imaging.
  Interventions: Other: No intervention
- Glaucoma Cohort: Patients with glaucoma-related optic nerve damage undergoing OCT/OCTA imaging.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — This observational study involves no experimental intervention. All OCT and OCTA examinations are performed as part of routine clinical care, and the study only analyzes retrospectively and prospectively collected imaging and clinical data to evaluate a large-model-based AI diagnostic system.

SUMMARY:
This observational study aims to establish key technologies for high-throughput, large-model-based AI-assisted diagnosis using optical coherence tomography (OCT) and OCT angiography (OCTA). The study will collect real-world OCT/OCTA images and corresponding clinical information from patients with common blinding retinal and optic nerve diseases at Peking Union Medical College Hospital.

A high-throughput diagnostic framework based on large-scale artificial intelligence models will be developed and evaluated. The primary objective is to determine the diagnostic performance of the AI system, including its ability to identify diabetic retinopathy, branch retinal vein occlusion, central retinal vein occlusion, age-related macular degeneration, pathologic myopic choroidal neovascularization, and glaucoma-related optic nerve damage.

The results of this study are expected to support the development of standardized, efficient, and scalable AI-assisted diagnostic pathways for OCT imaging in clinical practice.

DETAILED DESCRIPTION:
This study investigates key technologies for high-throughput, large-model-based AI-assisted diagnosis using optical coherence tomography (OCT) and OCT angiography (OCTA). OCT/OCTA imaging has become an essential non-invasive tool for detecting and monitoring retinal and optic nerve diseases, yet manual interpretation remains time-consuming, experience-dependent, and limited by inter-observer variability. Recent advances in large artificial intelligence models provide an opportunity to develop scalable, generalizable diagnostic tools that can process large multimodal datasets and support clinical decision-making.

This observational study will enroll patients who undergo routine OCT and/or OCTA examinations at Peking Union Medical College Hospital and who are diagnosed with one or more of the following conditions: diabetic retinopathy, branch retinal vein occlusion, central retinal vein occlusion, age-related macular degeneration, pathologic myopic choroidal neovascularization, or glaucoma with optic nerve damage. The study will include both retrospectively collected and prospectively acquired imaging and clinical data, following standardized quality control and data-management procedures.

The high-throughput diagnostic framework will be trained and validated using large-scale image and clinical datasets. Primary outcomes include diagnostic performance metrics such as the area under the receiver operating characteristic curve (AUC). Secondary outcomes include sensitivity, specificity, and lesion-level or structural feature assessment when applicable. No experimental intervention will be introduced, and all imaging and clinical evaluations will follow standard clinical care.

The study aims to produce a robust, clinically relevant benchmark for large-model-based AI systems in OCT/OCTA interpretation and provide technical support for future integration of AI-assisted diagnostic tools into routine ophthalmic practice.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients of any age or sex who undergo OCT and/or OCT angiography (OCTA) examinations as part of routine clinical care at Peking Union Medical College Hospital.

  2. Clinical diagnosis of at least one of the following conditions: Diabetic retinopathy, Branch retinal vein occlusion, Central retinal vein occlusion, Age-related macular degeneration, Pathologic myopia with choroidal neovascularization and Glaucoma with optic nerve damage.

  3. Imaging quality sufficient for analysis based on predefined OCT/OCTA quality control criteria.

  4. Ability to provide informed consent (for prospective participants), or availability of medical records that meet institutional ethical requirements (for retrospective data).

Exclusion Criteria:

- 1. Poor-quality OCT/OCTA images that do not meet analysis standards (e.g., severe motion artifacts, media opacity, incomplete scans).

2. Patients unable to cooperate with standard ophthalmic imaging procedures. 3. Any condition judged by investigators to preclude accurate imaging evaluation or reliable diagnostic interpretation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study population consists of patients who undergo OCT and/or OCT angiography (OCTA) examinations as part of routine clinical care at Peking Union Medical College Hospital. Eligible participants are clinically diagnosed with one or more of the following conditions: diabetic retinopathy, branch retinal vein occlusion, central retinal vein occlusion, age-related macular degeneration, pathologic myopia with choroidal neovascularization, or glaucoma with optic nerve damage. Both retrospectively collected and prospectively enrolled patients are included. No healthy volunteers or experimental interventions are involved.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2025-11-30 (Estimated); Primary Completion 2028-06-15 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic performance of the AI-assisted OCT/OCTA model (AUC for multi-disease classification) | Baseline imaging visit (time of image acquisition and model inference).
  Area under the receiver operating characteristic curve (AUC) of the high-throughput large-model-based OCT/OCTA diagnostic system for identifying major retinal and optic nerve diseases, including diabetic retinopathy, branch retinal vein occlusion, central retinal vein occlusion, age-related macular degeneration, pathologic myopic choroidal neovascularization, and glaucoma.

SECONDARY OUTCOMES:
Sensitivity and specificity of the AI-assisted OCT/OCTA model | At the time of image acquisition and model inference (baseline imaging visit).
  Sensitivity and specificity of the AI system for detecting each target disease (diabetic retinopathy, branch retinal vein occlusion, central retinal vein occlusion, age-related macular degeneration, pathologic myopic choroidal neovascularization, and glaucoma) compared with masked clinician consensus.
Agreement between AI-assisted diagnosis and clinician diagnosis | At the time of image acquisition and model inference (baseline imaging visit).
  Level of agreement between the AI system's classification and the final clinical diagnosis by retina and glaucoma specialists, quantified using Cohen's kappa statistics or similar agreement measures.

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data (IPD) are not planned for public sharing at this time due to institutional policies and ethical restrictions on releasing identifiable clinical imaging data. De-identified aggregated results may be shared upon reasonable request and in compliance with applicable regulations.